CLINICAL TRIAL: NCT00288639
Title: Lyrica (Pregabalin) Administered As An Add-On Therapy For Partial Seizures (LEADER) An Open-Label, Multicenter Add-On Therapy Trial
Brief Title: Lyrica (Pregabalin) Administered as an Add-on Therapy for Partial Seizures (LEADER).
Acronym: LEADER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081088
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2018-11

CONDITIONS: Epilepsy
Keywords: Pregabalin for partial seizures
MeSH Terms: conditions — Epilepsy | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pregabalin — Pregabalin treatment, given as 2 divided doses, is initiated at a dose of 150 mg/day (75 mg BID).
  Based on individual subject response and tolerability, the dosage may be increased to 300 mg/day after 1 week (150 mg BID given as two 75-mg capsules BID). Based on subjects individual response and tolerability, dosage can be incrementally increased further after an additional week to 600 mg/day (300 mg BID given as four 75-mg capsules BID).

SUMMARY:
The objective of study is to assess the clinical improvement (change in seizure frequency), safety, and tolerability of subjects with partial seizures following adjunctive therapy of pregabalin BID (150 to 600 mg/day titration) in addition to existing standards AEDs.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients equal to or greater than 18 years of age with diagnosis of epilepsy with partial seizures having minimum of two partial seizures during a two month period before the baseline visit
* Having a clinical history of epilepsy and AED treatment at least 1 year prior to inclusion

Exclusion Criteria:

* AED or Seizures/Epilepsy Related Exclusions:having a treatable cause of seizures
* Having absences seizures
* Having had status epileptics within the year prior to inclusion
* Having a progressive neurological or systematic disorder
* Having known significant renal or hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Greece (5):
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Heraklio
  - Pfizer Investigational Site, Mesogion, Athen
  - Pfizer Investigational Site, Pátrai
  - Pfizer Investigational Site, Thessaloniki

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081088&StudyName=Lyrica%20%28Pregabalin%29%20Administered%20in%20as%20an%20Add-on%20Therapy%20for%20Partial%20Seizures%20%28LEADER%29.%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned to enroll approximately 100 subjects with partial seizures at up to 10 study centers in Greece.
Pre-assignment Details: Single arm open label study without randomization. The study included the following 3 main phases with a total study treatment duration of up to 21 weeks: Treatment dose-optimization phase = 9 weeks. Treatment observation phase = 12 weeks.
Groups:
- Pregabalin: Pregabalin treatment, given as 2 divided doses, was initiated at a dose of 150 mg/day (75 mg BID). Then, based on individual subject response and tolerability, the dosage could have been increased to 300 mg/day after 1 week. The dosage could have been incrementally increased further to 600 mg/day after an additional week. After 9 weeks of treatment, the optimal dose of pregabalin was to be maintained for 3 months (12 week treatment observation period).
Period: Overall Study
Arm/Group | Pregabalin
Started | 98
Completed | 86
Not Completed | 12
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 98
Age, Customized [Number; unit: Participants]
  18 to 44 years | 69
  45 to 64 years | 25
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Partial Seizure Frequency (All Partial Seizure Types) Between Baseline and the 12 Week Observation Period
Description: Percentage change from baseline=[(12 week treatment observation period seizure frequency rate minus 8 week baseline period seizure frequency rate)/ 8 week baseline period seizure frequency rate] x 100. Seizure frequencies per 28-day period: = (total # of partial seizures in period x 28 / (total # of days in period).
Time Frame: 8 week baseline period & 12 week treatment observation period
Population: Full analysis set (FAS)/intent-to-treat (ITT) population (all subjects who received at least 1 dose of study treatment & had a minimum of 2 partial seizures during baseline period). Seizure rate was calculated on last observation carried forward (LOCF) basis, whereby data from last 84 days prior to last dose was used to calculate seizure frequency.
Measure: Median (Full Range); unit: percentage change in events
Arm/Group | Pregabalin
Number analyzed (Participants) | 92
percentage change in events | -33.33 [-100.00 to 7566.67]
Statistical Analysis 1: Comparison: Pregabalin; Noncomparative study. Summary stats, 2 sided 95% CI to est. effect size. No adjustments made to alpha levels to acct for multiple 2o endpts. Sample size=83 patients (pts) sufficient to detect statistically significant difference in % change from baseline in 28-day seizure rate with 80% power, true change from baseline approximately 25%. Allowing for dropouts assume 85% pts analyzed; Test type: Superiority or Other; Mean Response Ratio = -22.72, 95% CI [-34.16 to -11.28], Standard Deviation 55.232 — Response ratio = 100 x [(t - b)/(t + b)] where t=treatment seizure frequency and b=baseline seizure frequency

2. Secondary Outcome: Percentage Change in Partial Seizure Frequency (All Partial Seizure Types) Between Baseline and the Whole 21 Week Open-label Treatment Period.
Description: Percentage change from baseline = ((21 weeks-8 weeks)/8 weeks)*100. Negative mean R-Ratios and associated 95% CIs that do not include zero indicate reduction in partial seizure frequency.
Time Frame: 8 week baseline period and 21 week treatment period
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage change in events
Arm/Group | Pregabalin
Number analyzed (Participants) | 92
percentage change in events | -29.39 [-100.00 to 7478.95]
Statistical Analysis 1: Comparison: Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Response Ratio = -17.26, 95% CI [-27.36 to -7.15], Standard Deviation 48.797 — Response ratio = 100 x [(t - b)/(t + b)] where t=treatment seizure frequency and b=baseline seizure frequency

3. Secondary Outcome: Percentage Change in Partial Seizure Frequency (All Partial Seizure Types) Between the 8 Week Baseline Period and 4 Week Intervals During the 21 Week Open-label Treatment Period.
Description: Percentage change from baseline = [(4 week seizure frequency minus 8 week baseline) / (8 week baseline seizure frequency)] x 100. Negative mean R-Ratios and associated 95% CIs that do not include zero indicate reduction in partial seizure frequency.
Time Frame: 8 week baseline period and 21 week treatment period
Population: Full analysis set (FAS)/intent-to-treat (ITT) population (all subjects who received at least 1 dose of study treatment & had a minimum of 2 partial seizures during baseline period). Seizure date from patients who discontinued during any of these 4 week intervals will not be included in the summary for that interval.
Measure: Median (Full Range); unit: percentage change of events
Arm/Group | Pregabalin
Number analyzed (Participants) | 92
percentage change of events
  1-28 Days | -28.12 [-100.00 to 4833.33]
  29-56 Days | -22.50 [-100.00 to 9633.33]
  57-84 Days | -25.00 [-100.00 to 3433.33]
  85-112 Days | -40.00 [-100.00 to 5100.00]
  113-140 Days | -58.72 [-100.00 to 9166.67]
  >140 Days | -85.42 [-100.00 to 12344.44]
Statistical Analysis 1: Comparison: Pregabalin; Noncomparative study.Summary stats, 2 sided 95% CI to est. effect size. No adjustments made to alpha levels to acct for multiple 2o endpts.Sample size=83 patients (pts) sufficient to detect statistically significant difference in % change from baseline in 28-day seizure rate with 80% power, true change from baseline approximately 25%.Allowing for dropouts assume 85% pts analyzed; Test type: Superiority or Other; Mean Response Ratio = -22.43, 95% CI [-34.16 to -10.71], Standard Deviation 56.615 — 1-28 Days. Response ratio = 100 x [(t - b)/(t + b)] where t= 4 wk interval seizure frequency and b=baseline seizure frequency
Statistical Analysis 2: Comparison: Pregabalin; Noncomparative study.Summary stats, 2 sided 95% CI to est. effect size. No adjustments made to alpha levels to acct for multiple 2o endpts. Sample size=83 patients (pts) sufficient to detect statistically significant difference in % change from baseline in 28-day seizure rate with 80% power,true change from baseline approximately 25%. Allowing for dropouts assume 85% pts analyzed; Test type: Superiority or Other; Mean Response Ratio = -22.83, 95% CI [-34.74 to -10.91], Standard Deviation 57.543 — 29-56 Days. Response ratio = 100 x [(t - b)/(t + b)] where t= 4 wk interval seizure frequency and b=baseline seizure frequency
Statistical Analysis 3: Comparison: Pregabalin; Noncomparative study.Summary stats, 2 sided 95% CI to est. effect size. No adjustments made to alpha levels to acct for multiple 2o endpts. Sample size=83 patients (pts) sufficient to detect statistically significant difference in % change from baseline in 28-day seizure rate with 80% power, true change from baseline approximately 25%. Allowing for dropouts assume 85% pts analyzed; Test type: Superiority or Other; Mean Response Ratio = -27.18, 95% CI [-39.90 to -14.46], Standard Deviation 59.323 — 57-84 Days. Response ratio = 100 x [(t - b)/(t + b)] where t= 4 wk interval seizure frequency and b=baseline seizure frequency
Statistical Analysis 4: Comparison: Pregabalin; Noncomparative study.Summary stats, 2 sided 95% CI to est. effect size. No adjustments made to alpha levels to acct for multiple 2o endpts. Sample size=83 patients (pts) sufficient to detect statistically significant difference in % change from baseline in 28-day seizure rate with 80% power, true change from baseline approximately 25%.Allowing for dropouts assume 85% pts analyzed; Test type: Superiority or Other; Mean Response Ratio = -30.75, 95% CI [-43.44 to -18.06], Standard Deviation 58.110 — 85-112 Days. Response ratio=100 x [(t - b)/(t + b)] where t= 4 wk interval seizure frequency and b=baseline seizure frequency
Statistical Analysis 5: Comparison: Pregabalin; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; Mean Response Ratio = -38.75, 95% CI [-51.79 to -25.70], Standard Deviation 59.368 — 113-140 Days. Response ratio=100 x [(t - b)/(t + b)] where t= 4 wk interval seizure frequency and b=baseline seizure frequency
Statistical Analysis 6: Comparison: Pregabalin; Noncomparative study.Summary stats, 2 sided 95% CI to est. effect size. No adjustments made to alpha levels to acct for multiple 2o endpts. Sample size=83 patients (pts) sufficient to detect statistically significant difference in % change from baseline in 28-day seizure rate with 80% power,true change from baseline approximately 25%.Allowing for dropouts assume 85% pts analyzed; Test type: Superiority or Other; Mean Response Ratio = -44.24, 95% CI [-58.47 to -30.01], Standard Deviation 62.703 — >140 Days. Response ratio= 100 x [(t - b)/(t + b)] where t= 4 wk interval seizure frequency and b=baseline seizure frequency

4. Post Hoc Outcome: Change in Partial Seizure Frequency by Type Between the 8 Week Baseline Period and During the 12 Week Observation Period.
Description: Change from baseline = 12 week treatment observation period seizure frequency rate minus 8 week baseline period seizure frequency rate.
Time Frame: 8 week baseline period & 12 week treatment observation period
Population: as for outcome 1
Measure: Median (Full Range); unit: change in median partial seizures
Arm/Group | Pregabalin
Number analyzed (Participants) | 92
change in median partial seizures
  Simple Partial Seizures (n=47) | 0.00 [-15.50 to 149.67]
  Complex Partial Seizures (n=76) | 0.00 [-16.33 to 114.67]
  Evolve to Secondary Generalized (n=30) | 0.00 [-2.67 to 9.04]
Statistical Analysis 1: Comparison: Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Response Ratio = 7.19, 95% CI [-17.60 to 31.98], Standard Deviation 84.425 — Simple Partial Seizures. Response ratio = 100 x [(t - b)/(t + b)] where t=treatment seizure frequency and b=baseline seizure frequency
Statistical Analysis 2: Comparison: Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Response Ratio = -22.24, 95% CI [-37.80 to -6.69], Standard Deviation 68.058 — Complex Partial Seizures. Response ratio = 100 x [(t - b)/(t + b)] where t=treatment seizure frequency and b=baseline seizure frequency
Statistical Analysis 3: Comparison: Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Response Ratio = -23.85, 95% CI [-55.33 to 7.64], Standard Deviation 84.313 — Evolved to Generalized. Response ratio = 100 x [(t - b)/(t + b)] where t=treatment seizure frequency and b=baseline seizure frequency

5. Secondary Outcome: Number of Subjects Seizure-free
Description: Count of subjects seizure free during the period.
Time Frame: last 4 weeks & whole 12 week treatment observation period
Population: Full analysis set(FAS)/intent-to-treat(ITT) all subjects who received >= 1 dose of study Tx & >= 2 partial seizures during baseline pd. LOCF if subjects withdrew then last 4 wks prior to last dose (but after visit 3). 12 wk subjects who withdrew were regarded as missing. n= # subjects evaluable for seizure freedom during defined observation pd.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 93
participants
  During 12 week Observation period (n=84) | 18
  During the last 4 weeks of Obs. period (n=86) | 30

6. Secondary Outcome: Reduction in Partial Seizure Frequency Between Baseline and the Final 4 Weeks of the Observation Period.
Description: Number of subjects with at least a 50% or 75% reduction in partial seizure frequency between baseline and treatment period.
Time Frame: 8 week baseline observation period & last 4 weeks of observation period
Population: Full analysis set (FAS)/intent-to-treat (ITT) population (all subjects who received at least 1 dose of study treatment & had a minimum of 2 partial seizures during baseline period). Patients who discontinued less than 4 weeks into the observation period (after Visit 3/week 9) will be regarded as missing. No data prior to week 9 will be used.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 93
participants
  >= 50% reduction | 42
  >= 75% reduction | 33

7. Secondary Outcome: Subjects Achieving Seizure Freedom During Observation Period
Description: Number of subjects achieving seizure freedom (no seizures) during last 4 weeks or duration of 12 week observation period.
Time Frame: Day 147 from the first dose of study drug
Population: Full analysis set (FAS)/intent-to-treat (ITT) population (all subjects who received at least 1 dose of study treatment & had a minimum of 2 partial seizures during baseline period).
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 93
participants
  seizure-free during last 4 weeks | 30
  seizure-free during 12 weeks | 18

8. Secondary Outcome: Change in Partial Seizure Frequency (All Partial Seizure Types) Between Baseline and the 12 Week Observation Period Categorized by Baseline Seizure Frequency
Description: Percentage change from baseline = ((12 weeks - 8 weeks)/8 weeks)*100. Negative mean R-Ratios and associated 95% CIs that do not include zero indicate reduction in partial seizure frequency.
Time Frame: 8 week baseline observation period & 12 week treatment observation period
Population: Full analysis set (FAS)/intent-to-treat (ITT) (all subjects who received at least 1 dose of study treatment & minimum 2 partial seizures during baseline pd). Seizure rate was calculated on last observation carried forward (LOCF) basis, whereby data from last 84 days prior to last dose was used to calculate seizure frequency.
Measure: Median (Full Range); unit: percentage change in events
Arm/Group | Pregabalin
Number analyzed (Participants) | 92
percentage change in events
  Baseline seizure frequency ≤3 per 28 days (n=43) | -33.33 [-100.00 to 7566.67]
  Baseline seizure frequency >3 per 28 days (n=49) | -21.99 [-100.00 to 516.09]
Statistical Analysis 1: Comparison: Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Response Ratio = -24.93, 95% CI [-43.66 to -6.20], Standard Deviation 60.867 — Seizure freq. ≤3 / 28 d. Resp. ratio = 100 x [(t - b)/(t + b)] where t=treatment seizure frequency and b=baseline seizure frequency
Statistical Analysis 2: Comparison: Pregabalin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Response Ratio = -20.78, 95% CI [-35.24 to -6.33], Standard Deviation 50.334 — Seizure freq. >3 / 28 d. Resp. ratio = 100 x [(t - b)/(t + b)] where t=treatment seizure frequency and b=baseline seizure frequency

9. Secondary Outcome: Impression of Change in Overall Status Using the Patient Global Impression of Change (PGIC)
Description: The PGIC is a patient-rated instrument that measures change in patient's overall status on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: End of 21-week treatment
Population: Full analysis set (FAS)/intent-to-treat (ITT) population (all subjects who received at least 1 dose of study treatment and had a minimum of 2 partial seizures during the baseline period).
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 93
participants
  Very Much Improved | 14
  Much Improved | 36
  Minimally Improved | 17
  No Change | 9
  Minimally Worse | 3
  Much Worse | 1
  Very Much Worse | 0
  Missing / Not Done | 13

10. Secondary Outcome: Subjects With Categorical Impression of Change in Overall Status Using the Clinical Global Impression of Change (CGIC)
Description: The CGIC is a clinician's judgment of the overall change in the patient's condition over a defined period on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: End of 21-week treatment
Population: as for outcome 9
Measure: Number; unit: partcipants
Arm/Group | Pregabalin
Number analyzed (Participants) | 93
partcipants
  Very Much Improved | 15
  Much Improved | 35
  Minimally Improved | 24
  No Change | 11
  Minimally Worse | 4
  Much Worse | 2
  Very Much Worse | 0
  Missing / Not Done | 2

11. Secondary Outcome: Changes From Baseline in Medical Outcomes Study (MOS) Sleep Scale Scores
Description: Subjects recall sleep related activities over the previous 4 weeks. Low scores reflect greater impairment (except sleep adequacy, optimal sleep, &quantity). Range = 0 - 100 for Sleep Disturbance, Snoring, Awaken Short of Breath, Sleep Adequacy, Somnolence, & Sleep Problems Index. Quantity of Sleep Range = 0 - 24. Optimal Sleep Range 0 - 1.
Time Frame: Baseline, end of 21-week treatment
Population: Full analysis set (FAS)/intent-to-treat (ITT) population (all subjects who received at least 1 dose of study treatment & had a minimum of 2 partial seizures during baseline period). "n" is the number of subjects contributing to the mean at the specified time point.
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 93
score on scale
  Sleep Disturbance (n=72) | -3.95 (20.787) [-8.83 to 0.94]
  Snoring (n=76) | 7.89 [1.97 to 13.82]
  Awaken Short of Breath (n=77) | -1.82 [-5.93 to 2.29]
  Quantity of Sleep (n=66) | 0.05 [-0.33 to 0.42]
  Sleep Adequacy (n=77) | 4.29 [-2.20 to 10.77]
  Somnolence (n=77) | 0.52 [-4.61 to 5.65]
  Sleep Problems Index (n=72) | -2.81 [-6.50 to 0.88]

12. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale(HADS) Depression and Anxiety Symptoms Subscales Between Baseline and Week 21.
Description: Change in total HADS score between Baseline and Week 21. Each of the 14 items is scored 0, 1, 2 or 3 where a score of 3 corresponds to the most anxious/depressed. 7-item depression and 7-item anxiety subscales are summed; each resulting in a total score of 0-21.
Time Frame: Baseline, End of 21-week treatment
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 93
score on scale
  HADS Depression Subscale (n=76) | -0.59 [-1.38 to 0.19]
  HADS Anxiety Subscale (n=76) | -1.68 [-2.60 to -0.76]

13. Secondary Outcome: Number of Subjects With a Weight Gain at End of Treatment of at Least 7% Relative to Baseline
Description: Count of subjects with a weight gain of at least 7 percent relative to baseline.
Time Frame: Baseline, End of 21-week treatment
Population: Safety population (all subjects who had taken at least
  1 dose of study drug).
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 98
participants
  Weight gain ≥7% to <10% | 8
  Weight gain ≥10% to <15% | 2
  Weight gain ≥15% to <20% | 2
  Weight gain ≥20% | 1

14. Secondary Outcome: Subjects Assessment of Optimal Sleep
Description: Number of subjects that responded optimal or non-optimal sleep in Optimal Sleep subscale of Medical Outcomes Study (MOS) Sleep scale.
Time Frame: Baseline, End of 21-week treatment
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 93
participants
  Optimal Sleep Baseline, Optimal Sleep Wk21 | 21
  Optimal Sleep Baseline, Non-Optimal Sleep Wk21 | 8
  Non-Optimal Sleep Baseline, Optimal Sleep Wk21 | 12
  Non-Optimal Sleep Baseline, Non-Optimal Sleep Wk21 | 25

ADVERSE EVENTS:
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 3
Other Adverse Events (participants affected / at risk) | 35
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pregabalin
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1/98
Balance Disorder (Nervous system disorders) | 1/98
Convulsion (Nervous system disorders) | 1/98
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pregabalin
Constipation (Gastrointestinal disorders) | 2/98
Asthenia (General disorders) | 2/98
Weight Increased (Investigations) | 3/98
Ataxia (Nervous system disorders) | 2/98
Convulsion (Nervous system disorders) | 4/98
Disturbance in Attention (Nervous system disorders) | 2/98
Dizziness (Nervous system disorders) | 5/98
Headache (Nervous system disorders) | 2/98
Somnolence (Nervous system disorders) | 20/98
Agitation (Psychiatric disorders) | 4/98
Gait Disturbance (General disorders) | 3/98
Oedema peripheral (General disorders) | 2/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.